CLINICAL TRIAL: NCT00000528
Title: Trials of Hypertension Prevention (TOHP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Model: Factorial | Purpose: Prevention
Other Study IDs: 47; U01HL037852 (NIH)
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2005-12

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension; Vascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension; Vascular Diseases | interventions — Diet; Clinical Trials, Phase III as Topic

INTERVENTIONS:
Behavioral: diet, sodium-restricted (Phase III) diet, sodium-restricted
Behavioral: diet, reducing (Phase III)

SUMMARY:
To determine if nonpharmacological interventions, including diet and lifestyle change, could prevent increases in arterial blood pressure leading to systemic hypertension.

DETAILED DESCRIPTION:
BACKGROUND:

High blood pressure affects between 15 and 30 percent of the adult population in the United States, and is a major contributor to some of the leading causes of death including coronary artery and cerebrovascular diseases. A substantial body of evidence from both population and laboratory studies indicates that a number of dietary and lifestyle factors are associated with the chronic and progressive increase in blood pressure with age, commonly observed in populations of industrialized countries. There are also an increasing number of reports of important reductions in blood pressure in persons with hypertension following treatment with a number of different non-pharmacological interventions. These observations have led to interest in the possibility of the primary prevention of hypertension through non-pharmacological intervention on factors related to the development of high blood pressure.

In 1979, the main results of the NHLBI-supported Hypertension Detection and Follow-up Program (HDFP), then the largest of the randomized clinical trials of antihypertensive drug treatment, were reported. This trial compared the effects of intensive systematic Stepped-Care drug treatment with Referred-Care in the community. These results confirmed findings of earlier and subsequently reported placebo-controlled trials that effective blood-pressure lowering in hypertensive individuals reduces the occurrence of stroke, congestive heart failure, and other complications of hypertension, and for the first time demonstrated a significant reduction of total mortality. The implications of the findings regarding recommendations for long-term drug treatment for tens of millions of Americans led several groups of investigators to consider alternative approaches to the control of hypertension. To the concerns of these clinicians about drug-related symptoms and economic costs were added additional questions regarding the safety of common antihypertensive agents in some hypertensive subgroups, based on the results of the Multiple Risk Factor Intervention Trial and on other evidence.

A number of small to moderate-sized randomized clinical trials of non-pharmacologic intervention in hypertension have been initiated during the past 5 years with NHLBI support. The Hypertension Prevention Trial (HPT) was the largest program studying the effectiveness of intervening in a non-hypertensive population. The HPT was a feasibility study to establish the ability to enroll in sufficient numbers men and women with diastolic blood pressure of 78-89 mm Hg; to determine if dietary intervention alone could achieve sustained weight reduction, and/or a decrease in sodium intake, or an increase in potassium intake along with sodium reduction in these subjects; and to study the effects of the interventions on blood pressure. If feasibility were demonstrated, the plan was to conduct a full-scale trial with incidence of frank hypertension as the outcome measure.

The HPT achieved its feasibility goals regarding recruitment of participants and weight reduction, but not for dietary sodium reduction and potassium increase. Some of the other dietary trials among non-hypertensive subjects have also achieved relatively small sodium changes (20-25 percent); a few have produced much larger changes, but only with short-term follow-up. Other experience has also shown that it is difficult to increase potassium intake by dietary means alone.

The importance of further work in this area has meanwhile been reinforced by conclusions of several expert groups convened by NHLBI. These have included the participants in the 1984 NIH Workshop on Nutrition and Hypertension and the 1984 Joint National Committee on Detection, Evaluation, and Treatment of High Blood Pressure, whose report addressed in some detail non-pharmacologic intervention and primary prevention.

DESIGN NARRATIVE:

Phase I was a pilot study to test the feasibility of providing and obtaining compliance with selected nutritional-behavioral, non-pharmacologic interventions and to measure the short-term effectiveness of the interventions on reducing or preventing an increase in diastolic blood pressure. Ten clinical centers, and a coordinating center, which included two central laboratories and a nutrient data center, participated. Each clinic tested a subset of the interventions. The lifestyle arm of the trial, which included weight loss, sodium restriction, and stress management, had an open design with untreated controls. The two-stage supplement arm of the trial, which tested magnesium and calcium in Stage I, and fish oil and potassium in Stage II, was double-blinded and placebo-controlled. Three clinics tested only lifestyle interventions, two tested only supplements, and five participated in both arms of the trial. Recruitment began in August 1987 and randomization was completed by October 1988. Endpoint data collection was completed in January 1990. The average follow-up was approximately 18 months.

Phase II had a 2x2 factorial design to test the effectiveness of weight loss and sodium restriction alone and in combination in reducing blood pressure and decreasing the incidence of definite hypertension. Lifestyle interventions were administered through counseling sessions at each center. Blood pressure, weight, body mass index, skin fold thickness, and urine electrolytes were measured at baseline and at six month intervals for a minimum of 36 months. Recruitment began at the end of 1990 and was completed in March 1992. Intervention and follow-up were completed in March 1995. Data analysis continued through June 1998 under U01-HL-37852, the coordinating center.

The main results were presented at the 1995 American Heart Association Scientific Sessions. The Phase II main results paper was published in March 1997.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
Men and women, ages 30 to 54, with high normal diastolic blood pressure between 83 and 89 mm Hg.

Subjects were mildly obese.

Ages: 30 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1986-09; Study Completion 1998-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Hennekens — Brigham and Women's Hospital

REFERENCES:
- [Background] Kumanyika SK, Obarzanek E, Stevens VJ, Hebert PR, Whelton PK, Kumanyaka SK. Weight-loss experience of black and white participants in NHLBI-sponsored clinical trials. Am J Clin Nutr. 1991 Jun;53(6 Suppl):1631S-1638S. doi: 10.1093/ajcn/53.6.1631S. PMID 2031498
- [Background] Rosner B, Langford HG. Judging the effectiveness of antihypertensive therapy in an individual patient. J Clin Epidemiol. 1991;44(8):831-8. doi: 10.1016/0895-4356(91)90138-y. PMID 1941036
- [Background] Whelton PK, Hebert PR, Cutler J, Applegate WB, Eberlein KA, Klag MJ, Keough ME, Hamill S, Borhani NO, Hollis J, et al. Baseline characteristics of participants in phase I of the Trials of Hypertension Prevention. Ann Epidemiol. 1992 May;2(3):295-310. doi: 10.1016/1047-2797(92)90062-u. PMID 1342280
- [Background] The effects of nonpharmacologic interventions on blood pressure of persons with high normal levels. Results of the Trials of Hypertension Prevention, Phase I. JAMA. 1992 Mar 4;267(9):1213-20. doi: 10.1001/jama.1992.03480090061028. PMID 1586398
- [Background] Kumanyika SK, Hebert PR, Cutler JA, Lasser VI, Sugars CP, Steffen-Batey L, Brewer AA, Cameron M, Shepek LD, Cook NR, et al. Feasibility and efficacy of sodium reduction in the Trials of Hypertension Prevention, phase I. Trials of Hypertension Prevention Collaborative Research Group. Hypertension. 1993 Oct;22(4):502-12. doi: 10.1161/01.hyp.22.4.502. PMID 8406655
- [Background] Satterfield S, Borhani NO, Whelton P, Goodwin L, Brinkmann C, Charleston J, Corkery BW, Dolan L, Hataway H, Hertert S, et al. Recruitment for phase I of the trials of hypertension prevention. Am J Prev Med. 1993 Jul-Aug;9(4):237-43. PMID 8398224
- [Background] Cook NR, Rosner BA. Screening rules for determining blood pressure status in clinical trials. Application to the trials of hypertension prevention. Am J Epidemiol. 1993 Jun 15;137(12):1341-52. doi: 10.1093/oxfordjournals.aje.a116643. PMID 8333415
- [Background] Stevens VJ, Corrigan SA, Obarzanek E, Bernauer E, Cook NR, Hebert P, Mattfeldt-Beman M, Oberman A, Sugars C, Dalcin AT, et al. Weight loss intervention in phase 1 of the Trials of Hypertension Prevention. The TOHP Collaborative Research Group. Arch Intern Med. 1993 Apr 12;153(7):849-58. PMID 8466377
- [Background] Kahn HA, Whelton PK, Appel LJ, Kumanyika SK, Meneses JL, Hebert PR, Woods M. Validity of 24-hour dietary recall interviews conducted among volunteers in an adult working community. Ann Epidemiol. 1995 Nov;5(6):484-9. doi: 10.1016/1047-2797(95)00065-8. PMID 8680612
- [Background] Appel LJ, Hebert PR, Cohen JD, Obarzanek E, Yamamoto M, Buring J, Stevens V, Kirchner K, Borhani NO. Baseline characteristics of participants in phase II of the Trials of Hypertension Prevention (TOHP II). Trials of Hypertension Prevention (TOHP) Collaborative Research Group. Ann Epidemiol. 1995 Mar;5(2):149-55. doi: 10.1016/1047-2797(94)00059-3. PMID 7795833
- [Background] Whelton PK, Buring J, Borhani NO, Cohen JD, Cook N, Cutler JA, Kiley JE, Kuller LH, Satterfield S, Sacks FM, et al. The effect of potassium supplementation in persons with a high-normal blood pressure. Results from phase I of the Trials of Hypertension Prevention (TOHP). Trials of Hypertension Prevention (TOHP) Collaborative Research Group. Ann Epidemiol. 1995 Mar;5(2):85-95. doi: 10.1016/1047-2797(94)00053-v. PMID 7795836
- [Background] Yamamoto ME, Applegate WB, Klag MJ, Borhani NO, Cohen JD, Kirchner KA, Lakatos E, Sacks FM, Taylor JO, Hennekens CH. Lack of blood pressure effect with calcium and magnesium supplementation in adults with high-normal blood pressure. Results from Phase I of the Trials of Hypertension Prevention (TOHP). Trials of Hypertension Prevention (TOHP) Collaborative Research Group. Ann Epidemiol. 1995 Mar;5(2):96-107. doi: 10.1016/1047-2797(94)00054-w. PMID 7795837
- [Background] Hebert PR, Bolt RJ, Borhani NO, Cook NR, Cohen JD, Cutler JA, Hollis JF, Kuller LH, Lasser NL, Oberman A, et al. Design of a multicenter trial to evaluate long-term life-style intervention in adults with high-normal blood pressure levels. Trials of Hypertension Prevention (phase II). Trials of Hypertension Prevention (TOHP) Collaborative Research Group. Ann Epidemiol. 1995 Mar;5(2):130-9. doi: 10.1016/1047-2797(94)00057-z. PMID 7795831
- [Background] Lasser VI, Raczynski JM, Stevens VJ, Mattfeldt-Beman MK, Kumanyika S, Evans M, Danielson E, Dalcin A, Batey DM, Belden LK, et al. Trials of Hypertension Prevention, phase II. Structure and content of the weight loss and dietary sodium reduction interventions. Trials of Hypertension Prevention (TOHP) Collaborative Research Group. Ann Epidemiol. 1995 Mar;5(2):156-64. doi: 10.1016/1047-2797(94)00060-7. PMID 7795834
- [Background] Cook NR, Cohen J, Hebert PR, Taylor JO, Hennekens CH. Implications of small reductions in diastolic blood pressure for primary prevention. Arch Intern Med. 1995 Apr 10;155(7):701-9. PMID 7695458
- [Background] Whelton PK, Kumanyika SK, Cook NR, Cutler JA, Borhani NO, Hennekens CH, Kuller LH, Langford H, Jones DW, Satterfield S, Lasser NL, Cohen JD. Efficacy of nonpharmacologic interventions in adults with high-normal blood pressure: results from phase 1 of the Trials of Hypertension Prevention. Trials of Hypertension Prevention Collaborative Research Group. Am J Clin Nutr. 1997 Feb;65(2 Suppl):652S-660S. doi: 10.1093/ajcn/65.2.652S. PMID 9022561
- [Background] Effects of weight loss and sodium reduction intervention on blood pressure and hypertension incidence in overweight people with high-normal blood pressure. The Trials of Hypertension Prevention, phase II. The Trials of Hypertension Prevention Collaborative Research Group. Arch Intern Med. 1997 Mar 24;157(6):657-67. PMID 9080920
- [Background] Pickering TG. Lessons from the Trials of Hypertension Prevention, phase II. Energy intake is more important than dietary sodium in the prevention of hypertension. Arch Intern Med. 1997 Mar 24;157(6):596-7. No abstract available. PMID 9080913
- [Background] Hunt SC, Cook NR, Oberman A, Cutler JA, Hennekens CH, Allender PS, Walker WG, Whelton PK, Williams RR. Angiotensinogen genotype, sodium reduction, weight loss, and prevention of hypertension: trials of hypertension prevention, phase II. Hypertension. 1998 Sep;32(3):393-401. doi: 10.1161/01.hyp.32.3.393. PMID 9740601
- [Background] Kotchen TA. Angiotensinogen genotype and blood pressure responses to reduced dietary NaCl and to weight loss. Hypertension. 1998 Sep;32(3):402-3. doi: 10.1161/01.hyp.32.3.402. No abstract available. PMID 9740602
- [Background] Cook NR, Kumanyika SK, Cutler JA. Effect of change in sodium excretion on change in blood pressure corrected for measurement error. The Trials of Hypertension Prevention, Phase I. Am J Epidemiol. 1998 Sep 1;148(5):431-44. doi: 10.1093/oxfordjournals.aje.a009668. PMID 9737555
- [Background] Cook NR. An imputation method for non-ignorable missing data in studies of blood pressure. Stat Med. 1997 Dec 15;16(23):2713-28. doi: 10.1002/(sici)1097-0258(19971215)16:233.0.co;2-s. PMID 9421871
- [Background] Batey DM, Kaufmann PG, Raczynski JM, Hollis JF, Murphy JK, Rosner B, Corrigan SA, Rappaport NB, Danielson EM, Lasser NL, Kuhn CM. Stress management intervention for primary prevention of hypertension: detailed results from Phase I of Trials of Hypertension Prevention (TOHP-I). Ann Epidemiol. 2000 Jan;10(1):45-58. doi: 10.1016/s1047-2797(99)00041-1. PMID 10658688
- [Background] Hollis JF, Satterfield S, Smith F, Fouad M, Allender PS, Borhani N, Charleston J, Hirlinger M, King N, Schultz R, et al. Recruitment for phase II of the Trials of Hypertension Prevention. Effective strategies and predictors of randomization. Trials of Hypertension Prevention (TOHP) Collaborative Research Group. Ann Epidemiol. 1995 Mar;5(2):140-8. doi: 10.1016/1047-2797(94)00058-2. PMID 7795832
- [Background] Stevens VJ, Obarzanek E, Cook NR, Lee IM, Appel LJ, Smith West D, Milas NC, Mattfeldt-Beman M, Belden L, Bragg C, Millstone M, Raczynski J, Brewer A, Singh B, Cohen J; Trials for the Hypertension Prevention Research Group. Long-term weight loss and changes in blood pressure: results of the Trials of Hypertension Prevention, phase II. Ann Intern Med. 2001 Jan 2;134(1):1-11. doi: 10.7326/0003-4819-134-1-200101020-00007. PMID 11187414
- [Background] Kumanyika SK, Cook NR, Cutler JA, Belden L, Brewer A, Cohen JD, Hebert PR, Lasser VI, Raines J, Raczynski J, Shepek L, Diller L, Whelton PK, Yamamoto M; Trials of Hypertension Prevention Collaborative Research Group. Sodium reduction for hypertension prevention in overweight adults: further results from the Trials of Hypertension Prevention Phase II. J Hum Hypertens. 2005 Jan;19(1):33-45. doi: 10.1038/sj.jhh.1001774. PMID 15372064
- [Background] Cook NR, Kumanyika SK, Cutler JA, Whelton PK; Trials of Hypertension Prevention Collaborative Research Group. Dose-response of sodium excretion and blood pressure change among overweight, nonhypertensive adults in a 3-year dietary intervention study. J Hum Hypertens. 2005 Jan;19(1):47-54. doi: 10.1038/sj.jhh.1001775. PMID 15343354
- [Background] Satterfield S, Cutler JA, Langford HG, Applegate WB, Borhani NO, Brittain E, Cohen JD, Kuller LH, Lasser NL, Oberman A, et al. Trials of hypertension prevention. Phase I design. Ann Epidemiol. 1991 Aug;1(5):455-71. doi: 10.1016/1047-2797(91)90014-4. PMID 1669525
- [Background] Sacks FM, Hebert P, Appel LJ, Borhani NO, Applegate WB, Cohen JD, Cutler JA, Kirchner KA, Kuller LH, Roth KJ, et al. Short report: the effect of fish oil on blood pressure and high-density lipoprotein-cholesterol levels in phase I of the Trials of Hypertension Prevention. J Hypertens. 1994 Feb;12(2):209-13. PMID 8021472
- [Background] Sacks FM, Hebert P, Appel LJ, Borhani NO, Applegate WB, Cohen JD, Cutler JA, Kirchner KA, Kuller LH, Roth KJ, et al. The effect of fish oil on blood pressure and high-density lipoprotein-cholesterol levels in phase I of the Trials of Hypertension Prevention. Trials of Hypertension Prevention Collaborative Research Group. J Hypertens Suppl. 1994;12(7):S23-31. PMID 7769501